CLINICAL TRIAL: NCT05100303
Title: An Open-label, Multi-center Phase Ib/II Study to Evaluate the Tolerance and Efficacy of Mitoxantrone Hydrochloride Liposome Injection Combined With Cytarabine in Patients With Acute Myeloid Leukemia (AML)
Brief Title: A Study to Evaluate the Tolerance and Efficacy of Mitoxantrone Hydrochloride Liposome Injection Combined With Cytarabine in Patients With Acute Myeloid Leukemia (AML)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE071-CSP-022
Record Dates: First submitted 2021-10-19; First posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Treatment-naive or Relapsed or Refractory Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute | interventions — Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mitoxantrone Hydrochloride liposome and cytarabine (Experimental): Chemotherapy will be given in 28-day cycles, and total treatment period is 2 cycles.
  Dose escalation phase:
  Patients will receive 24 mg/m^2, 30 mg/m^2 or 36mg/m^2 of mitoxantrone hydrochloride liposome daily by intravenous (IV) injections on the first day and 1.5 g/m^2 of cytarabine twice daily by IV for 3 days (day 1, day3 and day5).
  Dose expansion phase:
  Patients with newly diagnosed AML will receive mitoxantrone hydrochloride liposome daily by IV on the first day, 100~200 mg/m^2 of cytarabine by IV for 7 days (day 1~7). Patients with R/R AML will receive mitoxantrone hydrochloride liposome daily by IV on the first day, 1.5 g/m^2 of cytarabine twice daily by IV for 3 days (day 1, day3 and day5). The dose size of mitoxantrone hydrochloride liposome will be determined by the investigator and the sponsor based on the results of the previous study.
  Interventions: Drug: Mitoxantrone Hydrochloride liposome injection; Drug: Cytarabine (LoDAC)

INTERVENTIONS:
Drug: Mitoxantrone Hydrochloride liposome injection — Mitoxantrone hydrochloride liposome will be administered by intravenous (IV) injections.
Drug: Cytarabine (LoDAC) — Low-dose or high-dose cytarabine (LoDAC) will be administered by intravenous (IV) injections.

SUMMARY:
This is an open-label, multi-cohort, multi-center Phase Ib/II clinical study to evaluate the tolerance and efficacy of Mitoxantrone Hydrochloride liposome injection combined with cytarabine in patients with Acute Myeloid Leukemia (AML). The study will be divided into two phases, the dose escalation phase and the dose expansion phase. Patients with relapsed or refractory(R/R) AML will be included in the dose-escalation phase, and patients with treatment-naïve or R/R AML will be included in the dose-expansion phase.

DETAILED DESCRIPTION:
Dose escalation phase: Eligible patients will enter the screening period up to 14 days before the start of treatment. Patients will receive mitoxantrone liposomes combined with cytarabine, with a fixed dose of cytarabine and mitoxantrone liposomes in 3 dose groups: 24 mg/m^2, 30 mg/m^2 and 36 mg/m^2. The starting dose will be 24 mg/m^2, and the "3+3" principle is adopted for the escalation. If the maximum tolerated dose is not explored at the preset maximum dose (36 mg/m^2), the investigator and the sponsor will determine whether to continue the dose escalation, and it is necessary to ensure that 6 patients complete the dose-limiting toxicity (DLT) observation under this dose group. The treatment period includes 2 cycles with each cycle lasting 28 days. Cycle 1 is the DLT observation period and Cycle 2 is the extended dosing period. Mitoxantrone hydrochloride liposome injection will be given on the first day of each cycle, and cytarabine will be given every 12 hours on Day 1, 3, and 5 of each cycle. Patients who do not experience a DLT in the first cycle and achieve is at least PR, may enter the extended dosing period and be treated with the original regimen in Cycle 2. Patients who have completed 2 cycles and have a DLT in the first cycle or have not achieved PR will be withdrawn from treatment.

Dose expansion phase: Newly treated AML or R/R AML patients will be included and divided into two cohorts. Eligible patients will enter the screening period up to 14 days before receiving treatments. The treatment period is 2 cycles, and each cycle is 28 days. Mitoxantrone hydrochloride liposome injection will be given on the first day of each cycle, whose dose size will be determined by the investigator and the sponsor based on the results of the previous study. Cytarabine will be given on Day 1-7 of each cycle for the treatment-naïve group, and on Day 1, 3 and 5 of each cycle for the R/R group. Patients will take 1 cycle of therapy and will be assessed for response at the end of the 1st cycle. After the efficacy evaluation, the patient may receive a second cycle of chemotherapy at the investigator's discretion. And patients whose curative effect do not reach PR will be withdrawn from treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients volunteer to participate in this study and sign the informed consent form.
2. Age≥18 years old, no gender limitation.
3. Patient has a diagnosis of newly diagnosed or relapsed or refractory(R/R) AML as determined by pathological and morphological results, according to World Health Organization (WHO) 2016 classification.
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
5. Patient must meet the following criteria as indicated on the clinical laboratory tests:a. Serum aspartate aminotransferase and alanine aminotransferase ≤ 3.0 x upper limit of normal (ULN);b. Serum total bilirubin ≤ 1.5 x ULN;c. Serum creatinine ≤ 1.5 x ULN.
6. Patient and their partner agree to take effective contraception from the date of signing an informed consent to 180 days after the last dose; female patients must have negative urine or blood HCG (except for menopause and hysterectomy).

Exclusion Criteria:

1. Any of the following cases:(1) diagnosed as acute promyelocytic leukemia (APL);(2) chronic myelogenous leukemia in blast crisis;(3) AML with central nervous system leukemia.
2. Patient has been previously diagnosed with another malignancy in last 5 years (except for cured basal cell carcinoma of skin or cervical carcinoma in situ).
3. Patient is receiving continuous treatment for graft-versus-host disease (GVHD), or has received autologous or allogeneic stem cell transplantation more than once.
4. Allergic history of mitoxantrone hydrochloride injection, cytarabine or liposome.
5. Previously received doxorubicin or other anthracyclines, and the cumulative dose of doxorubicin exceeds 400 mg/m^2 (calculation of equivalent dose of anthracyclines: 1 mg doxorubicin = 2 mg epirubicin = 2 mg daunorubicin = 0.5 mg noroxydaunorubicin = 0.45 mg mitoxantrone; except doxorubicin liposomes).
6. Patient has received any anti-tumor treatment within 2 weeks before the first dose (or within 5 half-lives of the drug), including chemotherapy, immunotherapy, targeted therapy, endocrine therapy and radiation therapy (local radiation therapy interval < 2 weeks). Leukopenia treatment (hydroxyurea, leukocyte separation, etc.) and preventive intrathecal injection exceeds 24 hours are the exception.
7. The non-hematological toxicity of previous anti-tumor treatment does not return to grade≤1 (except for alopecia, skin pigmentation or tolerable events judged by the investigator).
8. Patient is receiving systemic anti-infection treatment but has poor response (there are signs of infection progression within 1 week prior to the first dose or determined by the investigator).
9. The estimated survival time is less than 3 months.
10. Any of the following conditions occurs in cardiac function:(1) Long QTc syndrome or QTc interval > 480 ms;(2) Complete left bundle branch block or severe atrioventricular block disease (except for patients who use the pacemaker);(3) Serious and uncontrolled arrhythmias and unstable angina pectoris requiring drug treatment;(4) History of chronic congestive heart failure, New York Heart Association (NYHA)≥grade 3;(5) The cardiac ejection fraction is less than 50% or lower than the lower limit of the laboratory test value range of the research center;(6)Uncontrollable hypertension (defined as multiple measurements of systolic blood pressure > 150 mmHg or diastolic blood pressure > 90 mmHg under drug control);(7) History of myocardial infarction, unstable angina pectoris, viral myocarditis or severe pericardial disease, ECG evidence of acute ischemia or active conduction system abnormalities within 6 months before screening.
11. Patients have thromboembolic events in the past 6 months, such as cerebrovascular accidents (including transient ischemic attack) and pulmonary embolism.
12. HBsAg/HBcAb positive with HBV-DNA ≥2000 IU/mL, hepatitis C antibody-positive with HCV-RNA higher than the lower limit of the detection value of the research center, or HIV antibody positive in the preliminary screening.
13. Patients who have undergone major surgery (except intravenous infusion port implantation) within 3 months before the first study dose, or plan to perform major surgery during the study period.
14. Patient is suffering from any serious and /or non-controllable disease, or the investigator determines that the disease might affect the participants in the study, including (but not limited to, uncontrolled diabetes, dialysis related kidney diseases, severe liver diseases, life-threatening autoimmune diseases and hemorrhagic diseases, drug abuse, neurological diseases, etc.).
15. Pregnant or lactating female.
16. Patients are not suitable for the study in the investigator's opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Occurrence of dose-limiting toxicity (DLT)in dose escalation phase | The first cycle (28 days)
Adverse events during treatment in dose expansion phase | up to 3 years

SECONDARY OUTCOMES:
Adverse events during treatment in dose escalation phase | up to 3 years
Composite CR rate (CRc: CR+CRi) in dose escalation phase | up to 3 years
Objective response rate (ORR) in dose escalation phase | up to 3 years
Overall survival (OS) in dose escalation phase | up to 3 years
Explore maximum tolerated dose (MTD) in dose escalation phase | up to 3 years
Composite CR rate (CRc: CR+CRi) in dose expansion phase | up to 3 years
Objective response rate (ORR) in dose expansion phase | up to 3 years
Overall survival (OS) in dose expansion phase | up to 3 years
Explore RP2D in dose expansion phase | up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou, China